CLINICAL TRIAL: NCT06366061
Title: A COMPARISON OF LEFT VENTRICULAR FUNCTION IN THE APICAL 4 CHAMBER AND SUBCOSTAL 4 CHAMBER TTE VIEWS IN THE PERIOPERATIVE SETTING: A PROSPECTIVE, CLINICAL TRIAL
Brief Title: A COMPARISON OF LEFT VENTRICULAR FUNCTION IN THE APICAL 4 CHAMBER AND SUBCOSTAL 4 CHAMBER TTE VIEWS IN THE PERIOPERATIVE SETTING
Status: Recruiting | Type: Observational
Sponsor: Eckhard Mauermann (Other)
Responsible Party: Sponsor-Investigator, Eckhard Mauermann, PD, University Hospital, Basel, Switzerland
Organization: University Hospital, Basel, Switzerland (Other)
Other Study IDs: 2020-02868
Record Dates: First submitted 2022-05-13; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Cardiac Functional Disturbances During Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Randomization: A randomization will be done for the order of the different TTE measurments, but all patients are going the same TTE measurements after all

SUMMARY:
This study aims to examine the correlation and agreement of regional and global measurements of ventricular function in the apical 4 chamber and subcostal 4 chamber view. Additionally, we will explore limitations of the technology and explore the effect of left lateral positioning.

DETAILED DESCRIPTION:
In transthoracic echocardiography, a number of measures are endorsed by current guidelines for quantifying ventricular function. These include conventional (mitral annular plane velocities, ejection fraction) and novel, speckle-tracking (STE) technologies. However, these measurements are standardized to be measured in the left lateral decubitus position in the apical (4-chamber) view of awake spontaneously breathing patients.

In the perioperative period, however, attaining these measurements in the endorsed circumstances may be challenging for a number of reasons. First, obtaining usable AP4C images may be difficult in ventilated or post-surgical patients. While the SC4C is generally obtainable visualized structures are not identical to those of the AP4C and measurement technologies such as Doppler are misaligned Secondly, patient conditions (e.g. in distress, or during surgery) may preclude positioning the patient in the left lateral decubitus position. Finally, patients may be ventilated and under anesthesia.

Newer technologies - such as speckle-tracking- may partially overcome these difficulties as these technologies are considered to be relatively angle independent. For quantification, it would be important to know whether or not speckle-tracking based measurements in the SC4C are sufficiently close to those measured under the endorsed conditions.

ELIGIBILITY:
Inclusion Criteria:

* Consenting adult patients undergoing elective non-cardiac surgery

Exclusion Criteria:

* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Previous enrolment into the current study,
* Emergency procedures mandating expeditive patient care,
* Nonregular heart rhythm
* Valvular heart disease in the LV at least midgrade

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing elective non-cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-05-14 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
S'Tissue Doppler Index (TDI) AP4C supine vs. S'STE SC4C supine | This is going to be assessed after the trans thoracic echocardiography, through study completion (an average of 1 year)
  - Comparison of two velocities measured by two different methods.

SECONDARY OUTCOMES:
Global longitudinal strain (GLS), AP4C supine vs. GLS, SC4C supine, i.e. clinical questions: can we use the SC4C for global markers of ventricular function? | This is going to be assessed after the trans thoracic echocardiography, through study completion (an average of 1 year)
  * Correlation: GLS, AP4C, supine vs. GLS, SC4C supine
  * Bland Altman (BA) Plot: GLS, AP4C, supine vs. GLS, SC4C supine

OTHER OUTCOMES:
Comparison of high Frame Rate (FR) vs. low FR of the following measures: [ i) S'STE AP4C supine, ii) GLS AP4C supine, iii) SR AP4C supine] | This is going to be assessed after the trans thoracic echocardiography, through study completion (an average of 1 year)
  With high Frame Rate (FR) the measures will be more exact than with low FR
Comparison of the measured values in the cardiological gold standard (Left lateral decubitus (LLD)) vs. supine, for the following values [ i) S'TDI AP4C, ii) S'STE AP4C, iii) GLS] | This is going to be assessed after the trans thoracic echocardiography, through study completion (an average of 1 year)
  Comparison of values in different patient position for TTE

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No